CLINICAL TRIAL: NCT03821519
Title: Phase I/II Trial of Donor Derived Cytokine Induced Killer (CIK) Cells Infusion for Relapsed Hematologic Malignancy After Haploidentical Stem Cell Transplantation
Brief Title: Infusion of Donor Derived Cytokine Induced Killer (CIK) Cells in Hematological Patients Relapsed After Haploidentical Stem Cell Transplant
Acronym: Haplo-CIK
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Responsible Party: Principal Investigator, Rambaldi Alessandro, Head Hematology and Bone Marrow Transplant Unit, A.O. Ospedale Papa Giovanni XXIII
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2018-000716-24
Record Dates: First submitted 2019-01-22; First posted 2019-01-29 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Relapsed Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients relapse after haplo-HSCT for hematologic malignancies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Relapsed after Haplo transplant (Experimental)
  Interventions: Biological: donor-derived CIK cells

INTERVENTIONS:
Biological: donor-derived CIK cells — Treatment plan will be based on three infusions of donor derived CIK cells given by 3 weeks intervals at increasing dose levels. No dose changes are allowed and the following planned dose levels will be administered to each patient enrolled: 5x106, 5x106 and 10x106 cells/Kg according to the dose escalating program

SUMMARY:
The haematological neoplasia relapse is the cause of higher mortality after allogeneic stem cell transplantation (HSCT). When transplantation fails the most common therapeutic strategy is to increase the antitumor activity of the donor's immune system through the infusion of donor Lymphocytes (DLI). The use of DLI may limit the relapse, but may induce transplantation disease against the host (GvHD), in 40-60% of patients. With advances in transplantation procedures, the use of non-compatible (HLA-mismatched) haploidentical (aplo) donor cells has become feasible and is increasing. However, strategies for immune control of relapse after HSCT from haploidentical donor are hampered by the absence of prospective data that can guide treatment and limit the induction of GvHD in the setting of the HLA difference between the donor and the recipient. Cytokine-induced Killer Cells (CIK) are T lymphocytes from haploidentical donor expressing CD56 (e.g., double positive cells at CD3 / CD56). CIK are a product of advanced cell therapy (Advanced Therapeutic Medicinal Product, ATMP) for somatic cell therapy and have a reduced histocompatibility (MHC) complex: are cytotoxic, anti-tumor cells, possess the characteristics of both T cells and Natural Killer (NK) and show in vivo a very strong cytolytic activity against leukemia, but a low reactivity against the host. Therefore, this study has as its primary objective to investigate the safety of CIK cells deriving from the donor, especially in terms of the onset of GvHD, used as a treatment for relapse after transplantation with haploidentical stem cells. The study will allow to evaluate the possibility of using CIK cells, at the indicated dose combination (5x10 * 6 cells / kg, 5x10 * 6 and 10x10 * 6 cells / kg) as an effective and safe therapy in the context of haploidentical transplantation.

DETAILED DESCRIPTION:
Disease relapse is a major cause of mortality following allogeneic hematopoietic stem cell transplantation (HSCT) for hematologic malignancies. When allogeneic transplant fails the most common therapeutic strategy is to increase the anti-tumor activity of donor immune system through infusion of donor lymphocytes (DLI). Use of DLI can effectively treat limited relapses, but can induce graft-versus-host disease (GvHD) in the range of 40-60% of the patients. With the advances in HSCT procedure, the use of HLA-mismatched (haplo) family donors became feasible and extended the opportunity for HSCT to almost all patients lacking an HLA-matched donor. Due to the promising results of the procedure and the easier access to the donor, the number of haplo-HSCT transplant is steeply increasing. However, strategies aiming at eliciting the immune control of the relapse after haplo-HSCT are hampered by absence of prospective data that guide treatment and the fear of inducing GvHD in this setting of profound HLA disparity between donor and recipient.

* Despite the use of DLI in haplo-HSCT is not a standard practice, DLI are occasionally empirically used, mainly due to the lack of alternative treatment.
* Cytokine Induced Killer (CIK) cells are T lymphocytes expressing the CD56 marker, i.e. CIK are CD3/CD56 double positive cells. CIK cells are produced in vitro by incubating blood leukocytes according to a specific expansion protocol which includes initial stimulation with Interferon-gamma and anti-CD3 antibody, followed by expansion with (Interleukin-2) IL-2. CIK cells are non MHC restricted, cytotoxic, anti-tumoral cells which share characteristics of both T and NK cells and show in vivo a very strong cytolytic activity against leukemia, graft versus leukemia, while being essentially devoid of graft versus host reactivity. They show a natural non-MHC restricted (T Cell Receptor)TCR independent cytotoxicity against malignant targets cells, involving perforin and granzyme release and NKG2D, as well as CD56 and other small target molecules. In the past 15 years the investigators have extensively studied the use of cytokine-induced killer (CIK) cells as alternative cellular therapy to treat disease relapse after HSCT. The key feature of CIK cell therapy in the context of haplo- HSCT is the lower risk of inducing GvHD compared to DLI, that could permit to avoid the devastating effect of acute and chronic GvHD in terms of decreased survival, quality of life, disability and need of additional care. Indeed, beyond the dramatic impact in the quality and quantity of life of patients, costs for the health system of the management of acute and chronic GvHD are exceedingly high. At this regard, CIK cells have been regarded as the cellular therapy that is associated with a more favourable therapeutic index compared to DLI.
* In an early Phase I study the investigators observed remissions in 3 of 11 patients who were treated with infusion of CIK cells at a time when malignant cells were detectable. In each of these 3 cases, the patient had been previously treated unsuccessfully with conventional DLI. Successful remission induction by infusion of CIK cells after unsuccessful DLI suggests that the (Graft Versus Leukemia) GVL activity of CIK cells was attributable to NK-T cells. In a subsequent phase I clinical trial was assessed the feasibility of using CIK cells from HLA-matched sibling donors. Using a dose escalation design, the investigators showed that CIK cells could be given at doses as high as 1x10^8 per kg recipient body weight without causing acute infusion-related toxicity. The investigators recently reported the final results of a phase II multicenter pilot study, showing that CIK cell treatment for the relapse after HSCT is effective with a low toxicity in terms of GvHD compared to DLI. Importantly for the present proposal, in this study, 5 patients were treated in the context of haplo- HSCT. These did not show any different response or safety concern compared to other patients, suggesting the feasibility of this approach in a haploidentical context. Similarly, another study of CIK cellular therapy in HSCT including also patients with haploidentical donors confirmed the feasibility and safety of this approach. Considering that infused T cells are associated with risk of GvHD induction, especially in the haploidentical transplantation setting, novel cellular therapies manipulated to minimize GvHD while enhancing the graft-versus leukemia efficacy need to be tested in early phase clinical trials. Thus, the aim of the present proposal is to use CIK cells as a platform for a safe and effective cellular therapy in the context of haploidentical transplantation. As no dose limiting toxicity has been reached in phase I/II studies and no clear relationship among dose and both toxicity and response emerged so far, in the present study the investigators planned to use the final standard dose of our previous phase II study of 5x106 cells/kg, 5x10^6 and 10x10^6 cells/kg with no schedule modification . Three infusion of CIK cells will be administered every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 years or older
2. Patients treated with haploidentical allogeneic transplantation for hematologic malignancies, excluding Chronic Myeloid Leukemia (CML), such as acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), multiple myeloma (MM), myelofibrosis (MF) and myelodysplastic syndrome (MDS)
3. To be enrolled to the safety run-in cohort, patients must have:

   - Evidence of relapsed disease after allogeneic transplantation, including molecular, cytogenetic or overt hematologic relapse

   To be enrolled to the phase II cohort, patients must have:
   * Evidence of relapsed disease after allogeneic transplantation, including, molecular, cytogenetic or overt hematologic relapse, or
   * Mixed chimerism after the day +90, defined as <75% donor in unfractionated bone marrow and/or <75% donor in unfractionated Peripheral blood (PB) and/or <75% donor in fractionated CD3+ peripheral blood.
4. Availability of a donor willing to donate peripheral blood mononuclear cells
5. Withdrawn of immune suppression at least 3 weeks before the beginning of the cell therapy program
6. Written informed consent prior to any study procedures being performed
7. For female patients:

   1. being postmenopausal for at least 1 year before the screening visit,OR
   2. being surgically sterile, OR
   3. if they are of childbearing potential, must agree to practice highly effective method of contraception and one additional effective (barrier) method from the time of signing the informed consent until the end of study. Highly effective method of contraception includes: (i) combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, transdermal; (ii) progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, implantable (intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner, sexual abstinence) OR
   4. must agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject from the time of signing the informed consent until the end of study. [Periodic abstinence (eg, calendar, ovulation, symptothermal, postovulation methods), withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.]
8. For male patients, even if surgically sterilized (i.e., status postvasectomy): a) with female partners of childbearing potential: must agree to practice barrier contraception (condom with or without spermicide) from the time of signing the informed consent until the end of study and his female partner must agree to practice method of contraception including one of the following: estrogen and progestogen containing hormonal contraception; inhibition of ovulation: oral, intravaginal, transdermal; progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, implantable (intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion) from the time of signing the informed consent until the end of study.b) must agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject from the time of signing the informed consent until the end of study. [Periodic abstinence (eg, calendar, ovulation, symptothermal, postovulation methods), withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.] c) must agree to refrain from donating sperm

Exclusion Criteria:

The presence of any of the following will exclude a subject from study enrolment 1. Donors positive for HIV, (Hepatitis B virus) HBV, (Hepatitis C virus) HCV, Treponema or unfit to donate peripheral blood mononuclear cells 2. Patients with active grade 2 or more acute or moderate chronic GVHD at study entry or before CIK infusion 3. Patients with rapidly progressive disease or not controlled by palliative supportive treatments, including chemotherapy, and with life expectancy less than 8 weeks 4. Any serious medical or psychiatric illness, including drug or alcohol abuse, that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01-13 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Number of deaths related to study treatment death | Within 3 weeks after the last CIK cells infusion.
  Death, with related attributed cause of the event (e.g. treatment, toxicities, disease, other) will be assessed
Incidence of grade >=III acute GvHD | Within 3 weeks after the last CIK cells infusion.
  Will be collected: date of onset, organ involvement and maximum grade of acute GVHD Staging and Grading of Acute GvHD will be evaluated according to Glucksberg.
Incidence of grade >= III acute GvHD | at +100 days after the last infusion of CIK cells
  Will be collected: date of onset, organ involvement and maximum grade of acute GVHD. Staging and Grading of Acute GvHD will be evaluated according to Glucksberg.

SECONDARY OUTCOMES:
Incidence of any grade acute GvHD | at day +100 after last CIK infusion
  Will be collected: date of onset, organ involvement and maximum grade of acute GVHD. Staging and Grading of Acute GvHD will be evaluated according to Glucksberg criteria.
Incidence of any grade chronic GvHD | at days +100, +365 after last CIK infusion
  Chronic GVHD will be evaluated according to the National Institutes of Health
  Consensus Criteria for Clinical Trials in Chronic Graft-versus-Host Disease:
  Diagnosis and Staging Working Group Report. The following data will be collected: date of onset, organ involvement, maximum organ score and maximum global scoring of chronic GVHD.
Incidence of Adverse events (AEs) and laboratory abnormalities. | Up to 365 days from last CIK infusion
  Number, causality and intensity of all adverse events occurring during the study will be evaluated according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) V4.03 and MedDRA code (current version).
Evaluation of Response of Disease | at day +21, +100 and +365 after the last CIK cell infusion, or before if clinically indicated according to Investigator's judgment. For patients with acute leukemia disease response will be evaluated also after 60 days from the last CIK infusion.
  Response of Disease will be assessed based on detection of any evidence of molecular, cytogenetic, chimerism or hematologic disease progression, including loss of complete donor chimerism.
Progression Free Survival | Since enrollment up to 1 year after last cells infusion (day +365).
  Progression free survival will be estimated as the probability of patients of being alive free of progression (stable disease) or free of disease since enrollment up to
  1 year after last cells infusion (day +365). Thus, death for disease, disease relapse and disease progression are treated as events. (Death for other cause than disease will treated as competing events). Patients alive, patients in stable disease and those free of disease at their last follow-up will be censored.
Overall Survival | Since enrollment up to 365 days after last CIK infusion
  Overall survival will be estimated as the probability of survival irrespective of disease state since enrollment up to 1 year after last cells infusion (day +365).
  Patients alive at their last follow-up are censored.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Rambaldi, MD, Principal Investigator — A.O. Ospedale Papa Giovanni XXIII
Locations (1):
- A O Papa Giovanni XXIII, Bergamo, Italy

REFERENCES:
- [Background] Slavin S, Ackerstein A, Morecki S, Gelfand Y, Cividalli G. Immunotherapy of relapsed resistant chronic myelogenous leukemia post allogeneic bone marrow transplantation with alloantigen pulsed donor lymphocytes. Bone Marrow Transplant. 2001 Oct;28(8):795-8. doi: 10.1038/sj.bmt.1703223. PMID 11781634
- [Background] Ghiso A, Raiola AM, Gualandi F, Dominietto A, Varaldo R, Van Lint MT, Bregante S, Di Grazia C, Lamparelli T, Galaverna F, Stasia A, Luchetti S, Geroldi S, Grasso R, Colombo N, Bacigalupo A. DLI after haploidentical BMT with post-transplant CY. Bone Marrow Transplant. 2015 Jan;50(1):56-61. doi: 10.1038/bmt.2014.217. Epub 2014 Oct 13. PMID 25310304
- [Background] Franceschetti M, Pievani A, Borleri G, Vago L, Fleischhauer K, Golay J, Introna M. Cytokine-induced killer cells are terminally differentiated activated CD8 cytotoxic T-EMRA lymphocytes. Exp Hematol. 2009 May;37(5):616-628.e2. doi: 10.1016/j.exphem.2009.01.010. PMID 19375652
- [Background] de Lima M, Porter DL, Battiwalla M, Bishop MR, Giralt SA, Hardy NM, Kroger N, Wayne AS, Schmid C. Proceedings from the National Cancer Institute's Second International Workshop on the Biology, Prevention, and Treatment of Relapse After Hematopoietic Stem Cell Transplantation: part III. Prevention and treatment of relapse after allogeneic transplantation. Biol Blood Marrow Transplant. 2014 Jan;20(1):4-13. doi: 10.1016/j.bbmt.2013.08.012. Epub 2013 Sep 7. PMID 24018392
- [Background] Introna M, Borleri G, Conti E, Franceschetti M, Barbui AM, Broady R, Dander E, Gaipa G, D'Amico G, Biagi E, Parma M, Pogliani EM, Spinelli O, Baronciani D, Grassi A, Golay J, Barbui T, Biondi A, Rambaldi A. Repeated infusions of donor-derived cytokine-induced killer cells in patients relapsing after allogeneic stem cell transplantation: a phase I study. Haematologica. 2007 Jul;92(7):952-9. doi: 10.3324/haematol.11132. PMID 17606446
- [Background] Laport GG, Sheehan K, Baker J, Armstrong R, Wong RM, Lowsky R, Johnston LJ, Shizuru JA, Miklos D, Arai S, Benjamin JE, Weng WK, Negrin RS. Adoptive immunotherapy with cytokine-induced killer cells for patients with relapsed hematologic malignancies after allogeneic hematopoietic cell transplantation. Biol Blood Marrow Transplant. 2011 Nov;17(11):1679-87. doi: 10.1016/j.bbmt.2011.05.012. Epub 2011 May 25. PMID 21664472
- [Background] Introna M, Lussana F, Algarotti A, Gotti E, Valgardsdottir R, Mico C, Grassi A, Pavoni C, Ferrari ML, Delaini F, Todisco E, Cavattoni I, Deola S, Biagi E, Balduzzi A, Rovelli A, Parma M, Napolitano S, Sgroi G, Marrocco E, Perseghin P, Belotti D, Cabiati B, Gaipa G, Golay J, Biondi A, Rambaldi A. Phase II Study of Sequential Infusion of Donor Lymphocyte Infusion and Cytokine-Induced Killer Cells for Patients Relapsed after Allogeneic Hematopoietic Stem Cell Transplantation. Biol Blood Marrow Transplant. 2017 Dec;23(12):2070-2078. doi: 10.1016/j.bbmt.2017.07.005. Epub 2017 Jul 13. PMID 28712935
- [Background] Rettinger E, Huenecke S, Bonig H, Merker M, Jarisch A, Soerensen J, Willasch A, Bug G, Schulz A, Klingebiel T, Bader P. Interleukin-15-activated cytokine-induced killer cells may sustain remission in leukemia patients after allogeneic stem cell transplantation: feasibility, safety and first insights on efficacy. Haematologica. 2016 Apr;101(4):e153-6. doi: 10.3324/haematol.2015.138016. Epub 2016 Jan 14. No abstract available. PMID 26768688
- [Background] Cheson BD, Bennett JM, Kopecky KJ, Buchner T, Willman CL, Estey EH, Schiffer CA, Doehner H, Tallman MS, Lister TA, Lo-Coco F, Willemze R, Biondi A, Hiddemann W, Larson RA, Lowenberg B, Sanz MA, Head DR, Ohno R, Bloomfield CD; International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. Revised recommendations of the International Working Group for Diagnosis, Standardization of Response Criteria, Treatment Outcomes, and Reporting Standards for Therapeutic Trials in Acute Myeloid Leukemia. J Clin Oncol. 2003 Dec 15;21(24):4642-9. doi: 10.1200/JCO.2003.04.036. PMID 14673054
- [Background] Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA; Alliance, Australasian Leukaemia and Lymphoma Group; Eastern Cooperative Oncology Group; European Mantle Cell Lymphoma Consortium; Italian Lymphoma Foundation; European Organisation for Research; Treatment of Cancer/Dutch Hemato-Oncology Group; Grupo Espanol de Medula Osea; German High-Grade Lymphoma Study Group; German Hodgkin's Study Group; Japanese Lymphorra Study Group; Lymphoma Study Association; NCIC Clinical Trials Group; Nordic Lymphoma Study Group; Southwest Oncology Group; United Kingdom National Cancer Research Institute. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68. doi: 10.1200/JCO.2013.54.8800. PMID 25113753
- [Background] Cheson BD, Greenberg PL, Bennett JM, Lowenberg B, Wijermans PW, Nimer SD, Pinto A, Beran M, de Witte TM, Stone RM, Mittelman M, Sanz GF, Gore SD, Schiffer CA, Kantarjian H. Clinical application and proposal for modification of the International Working Group (IWG) response criteria in myelodysplasia. Blood. 2006 Jul 15;108(2):419-25. doi: 10.1182/blood-2005-10-4149. Epub 2006 Apr 11. PMID 16609072
- [Background] Dohner H, Estey E, Grimwade D, Amadori S, Appelbaum FR, Buchner T, Dombret H, Ebert BL, Fenaux P, Larson RA, Levine RL, Lo-Coco F, Naoe T, Niederwieser D, Ossenkoppele GJ, Sanz M, Sierra J, Tallman MS, Tien HF, Wei AH, Lowenberg B, Bloomfield CD. Diagnosis and management of AML in adults: 2017 ELN recommendations from an international expert panel. Blood. 2017 Jan 26;129(4):424-447. doi: 10.1182/blood-2016-08-733196. Epub 2016 Nov 28. PMID 27895058
- [Background] Kyle RA, Rajkumar SV. Criteria for diagnosis, staging, risk stratification and response assessment of multiple myeloma. Leukemia. 2009 Jan;23(1):3-9. doi: 10.1038/leu.2008.291. Epub 2008 Oct 30. PMID 18971951
- [Background] Tefferi A, Cervantes F, Mesa R, Passamonti F, Verstovsek S, Vannucchi AM, Gotlib J, Dupriez B, Pardanani A, Harrison C, Hoffman R, Gisslinger H, Kroger N, Thiele J, Barbui T, Barosi G. Revised response criteria for myelofibrosis: International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) and European LeukemiaNet (ELN) consensus report. Blood. 2013 Aug 22;122(8):1395-8. doi: 10.1182/blood-2013-03-488098. Epub 2013 Jul 9. PMID 23838352
- [Background] Kolb HJ. Graft-versus-leukemia effects of transplantation and donor lymphocytes. Blood. 2008 Dec 1;112(12):4371-83. doi: 10.1182/blood-2008-03-077974. PMID 19029455
- [Background] Marks DI, Lush R, Cavenagh J, Milligan DW, Schey S, Parker A, Clark FJ, Hunt L, Yin J, Fuller S, Vandenberghe E, Marsh J, Littlewood T, Smith GM, Culligan D, Hunter A, Chopra R, Davies A, Towlson K, Williams CD. The toxicity and efficacy of donor lymphocyte infusions given after reduced-intensity conditioning allogeneic stem cell transplantation. Blood. 2002 Nov 1;100(9):3108-14. doi: 10.1182/blood-2002-02-0506. PMID 12384406
- [Background] Tomblyn M, Lazarus HM. Donor lymphocyte infusions: the long and winding road: how should it be traveled? Bone Marrow Transplant. 2008 Nov;42(9):569-79. doi: 10.1038/bmt.2008.259. Epub 2008 Aug 18. PMID 18711351
- [Background] Dazzi F, Szydlo RM, Craddock C, Cross NC, Kaeda J, Chase A, Olavarria E, van Rhee F, Kanfer E, Apperley JF, Goldman JM. Comparison of single-dose and escalating-dose regimens of donor lymphocyte infusion for relapse after allografting for chronic myeloid leukemia. Blood. 2000 Jan 1;95(1):67-71. PMID 10607686
- [Background] Aversa F, Tabilio A, Velardi A, Cunningham I, Terenzi A, Falzetti F, Ruggeri L, Barbabietola G, Aristei C, Latini P, Reisner Y, Martelli MF. Treatment of high-risk acute leukemia with T-cell-depleted stem cells from related donors with one fully mismatched HLA haplotype. N Engl J Med. 1998 Oct 22;339(17):1186-93. doi: 10.1056/NEJM199810223391702. PMID 9780338
- [Background] Luznik L, O'Donnell PV, Symons HJ, Chen AR, Leffell MS, Zahurak M, Gooley TA, Piantadosi S, Kaup M, Ambinder RF, Huff CA, Matsui W, Bolanos-Meade J, Borrello I, Powell JD, Harrington E, Warnock S, Flowers M, Brodsky RA, Sandmaier BM, Storb RF, Jones RJ, Fuchs EJ. HLA-haploidentical bone marrow transplantation for hematologic malignancies using nonmyeloablative conditioning and high-dose, posttransplantation cyclophosphamide. Biol Blood Marrow Transplant. 2008 Jun;14(6):641-50. doi: 10.1016/j.bbmt.2008.03.005. PMID 18489989
- [Background] Passweg JR, Baldomero H, Bader P, Bonini C, Cesaro S, Dreger P, Duarte RF, Dufour C, Falkenburg JH, Farge-Bancel D, Gennery A, Kroger N, Lanza F, Nagler A, Sureda A, Mohty M; European Society for Blood and Marrow Transplantation (EBMT). Hematopoietic SCT in Europe 2013: recent trends in the use of alternative donors showing more haploidentical donors but fewer cord blood transplants. Bone Marrow Transplant. 2015 Apr;50(4):476-82. doi: 10.1038/bmt.2014.312. Epub 2015 Feb 2. PMID 25642761
- [Background] Yan CH, Liu DH, Xu LP, Liu KY, Zhao T, Wang Y, Chen H, Chen YH, Han W, Huang XJ. Modified donor lymphocyte infusion-associated acute graft-versus-host disease after haploidentical T-cell-replete hematopoietic stem cell transplantation: incidence and risk factors. Clin Transplant. 2012 Nov-Dec;26(6):868-76. doi: 10.1111/j.1399-0012.2012.01618.x. Epub 2012 Mar 20. PMID 22432715
- [Background] Zeidan AM, Forde PM, Symons H, Chen A, Smith BD, Pratz K, Carraway H, Gladstone DE, Fuchs EJ, Luznik L, Jones RJ, Bolanos-Meade J. HLA-haploidentical donor lymphocyte infusions for patients with relapsed hematologic malignancies after related HLA-haploidentical bone marrow transplantation. Biol Blood Marrow Transplant. 2014 Mar;20(3):314-8. doi: 10.1016/j.bbmt.2013.11.020. Epub 2013 Dec 1. PMID 24296490
- [Background] Goldsmith SR, Slade M, DiPersio JF, Westervelt P, Schroeder MA, Gao F, Romee R. Donor-lymphocyte infusion following haploidentical hematopoietic cell transplantation with peripheral blood stem cell grafts and PTCy. Bone Marrow Transplant. 2017 Dec;52(12):1623-1628. doi: 10.1038/bmt.2017.193. Epub 2017 Oct 16. PMID 29035393
- [Background] Rambaldi A, Biagi E, Bonini C, Biondi A, Introna M. Cell-based strategies to manage leukemia relapse: efficacy and feasibility of immunotherapy approaches. Leukemia. 2015 Jan;29(1):1-10. doi: 10.1038/leu.2014.189. Epub 2014 Jun 12. PMID 24919807